CLINICAL TRIAL: NCT03514173
Title: Analysis of Sociotechnical Acceptance and Workflow Integration of a Remote Patient Monitoring Device on an Intensive Care Unit
Brief Title: Staff Acceptance of Remote Patient Monitoring on Intensive Care Unit
Acronym: SARPI
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felix Balzer, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: SARPI
Record Dates: First submitted 2018-03-27; First posted 2018-05-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Remote Patient Monitoring on Intensive Care Unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Remote Patient Monitoring — Use of remote patient monitoring

SUMMARY:
The subject of the observation study with accompanying employee survey is the evaluation of a patient remote monitoring system (Vital Sync from Medtronic, hereinafter abbreviated as "Vital Sync") in intensive care medicine.

The aim of this research project is to determine whether the use of Vital Sync on an intensive care unit is accepted by medical and nursing staff and can be integrated into everyday work as an additional visualisation and analysis tool.

DETAILED DESCRIPTION:
In intensive care medicine, patient monitoring has become a standard that has led to a significant improvement in patient safety in recent decades. At the international level, minimum requirements for patient monitoring have been set out in guidelines and recommendations that represent milestones in patient safety, such as the Helsinki Declaration for Anaesthesiology and the Vienna Declaration for Intensive Care. With advances in digital health, there are new options for patient monitoring that may improve patient safety.

The concept of the Internet of Things has recently gained in importance. While the personal computer (PC) was long regarded as a prerequisite for making technologies accessible to people, the use of computer-supported electronic infrastructures has become ubiquitous. Today, more and more everyday devices are equipped with electronic circuits (microchip, memory chip), blurring earlier boundaries between hardware and software. In an intensive care unit - an environment with high operational reliability - ubiquitous computing means that the processing and visualization of medical data must not be limited to typical workstations at the patient's bedside. Instead, the accessibility of data relevant to medical decisions should result from clinical workflows, leading to the targeted provision of information as needed.

Although various remote patient monitoring systems from commercial providers are already available, little is known about how they can effectively support clinical processes. At the Charité, the working group "Data Science in Perioperative Care" of the Clinic for Anaesthesiology with focus on operative intensive care Charité - Universitätsmedizin Berlin, Campus Virchow and Campus Mitte is systematically evaluating the integration of such novel technologies with special consideration of the socio-technical dimension.

In the pre-implementation phase, 15 ICU staff members (physicians, nurses and respiratory therapists) will be involved into a semi-structured interview study. Results from this pre-implementation study will be validated via two independent surveys involving ICU staff members (n>100). In the post-implementation phase, two semi-structured interview studies will be conducted with key stakeholders of the ICU until data saturation is reached (n=5-10). The focus of this post-implementation interview studies will be to analyse the usability of the installed remote patient monitoring system as well as the success of the implementation and its contributing factors.

ELIGIBILITY:
Inclusion criteria:

From the Department for Anaesthesiology and operative Intensive Care, Charité - Universitätsmedizin Berlin, Campus Virchow- Klinikum and Campus Charité Mitte, Germany

* physicians
* specialist nurses
* respiratory therapists or respiratory therapists

Exclusion criteria:

* Rejection of participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From the Department for Anaesthesiology and operative Intensive Care, Charité - Universitätsmedizin Berlin, Campus Virchow- Klinikum and Campus Charité Mitte, Germany
  * physicians
  * specialist nurses
  * respiratory therapists or respiratory therapists
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptance of Remote Patient Monitoring Device on Intensive Care Unit | One year
  Acceptance of Remote Patient Monitoring Device (measured by the Likert scale on the question "What was the benefit of the new system for you?" 0=no benefit; 5=very high benefit)

SECONDARY OUTCOMES:
Structural Data of Intensive Care Unit | One year
  Number and arrangement of ICU beds (in numbers e.g. 1,2,3,4....)
Structural Data of Intensive Care Unit | One year
  utilization of ICU (in percent e.g. 50%, 40%...)
Structural Data of Intensive Care Unit | One year
  number of ventilated patients
Structural Data of Intensive Care Unit | One year
  care per patient ratio (nurse per patient, e.g. 1:1)
Structural Data of Intensive Care Unit | One year
  doctor per patient (doctor per patient, e.g. 1:1)
Structural Data of Intensive Care Unit | One year
  working hours of staff (e.g. 7am until 8pm)
Use of medical technology on Intensive Care Unit | One year
  emotions when using Vital Sync (on a Likert Scale 0=very annoyed, 5=very happy)
Use of medical technology on Intensive Care Unit | One year
  Usability (Validated by John Brooke in 1986: System User Scale using Likert Scales) (0=bad usability, 100=very good usability)
Usage of Vital Sync | One year
  usage time (in minutes) of Vital Sync (in min. per day)
Usage of Vital Sync | One year
  usage frequency of Vital Sync (e.g. x time per day)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Balzer, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin, Klinik für Anästhesiologie m.S. operative Intensivmedizin, Berlin, Germany

REFERENCES:
- [Derived] Balzer F, Agha-Mir-Salim L, Ziemert N, Schmieding M, Mosch L, Prendke M, Wunderlich MM, Memmert B, Spies C, Poncette AS. Staff perspectives on the influence of patient characteristics on alarm management in the intensive care unit: a cross-sectional survey study. BMC Health Serv Res. 2023 Jul 5;23(1):729. doi: 10.1186/s12913-023-09688-x. PMID 37407989
- [Derived] Mosch LK, Poncette AS, Spies C, Weber-Carstens S, Schieler M, Krampe H, Balzer F. Creation of an Evidence-Based Implementation Framework for Digital Health Technology in the Intensive Care Unit: Qualitative Study. JMIR Form Res. 2022 Apr 8;6(4):e22866. doi: 10.2196/22866. PMID 35394445
- [Derived] Poncette AS, Mosch LK, Stablo L, Spies C, Schieler M, Weber-Carstens S, Feufel MA, Balzer F. A Remote Patient-Monitoring System for Intensive Care Medicine: Mixed Methods Human-Centered Design and Usability Evaluation. JMIR Hum Factors. 2022 Mar 11;9(1):e30655. doi: 10.2196/30655. PMID 35275071
- [Derived] Poncette AS, Mosch L, Spies C, Schmieding M, Schiefenhovel F, Krampe H, Balzer F. Improvements in Patient Monitoring in the Intensive Care Unit: Survey Study. J Med Internet Res. 2020 Jun 19;22(6):e19091. doi: 10.2196/19091. PMID 32459655
- [Derived] Poncette AS, Spies C, Mosch L, Schieler M, Weber-Carstens S, Krampe H, Balzer F. Clinical Requirements of Future Patient Monitoring in the Intensive Care Unit: Qualitative Study. JMIR Med Inform. 2019 Apr 30;7(2):e13064. doi: 10.2196/13064. PMID 31038467